CLINICAL TRIAL: NCT05591157
Title: A Prospective Study for Evaluating the Safety and Performance of CSF-3 ECG Lead-I, HR and PR When Compared to ECG Holter
Brief Title: Evaluation of CSF-3 in Performing ECG
Acronym: ECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardiacSense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CSF-3 ECG
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Healthy; ECG
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: clinical study is a prospective, open, single-center study to evaluate the performance and accuracy of the ECG and heart rate calculation of the CSF-3 investigational Device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CSF-3 and ECG Holter (Experimental): At least 40 healthy subjects with no relevant or cardiac medical history and negative cardiac symptoms. Subjects will perform an ECG spot-check measurement using the CSF-3 Device while simultaneously being connected to an ECG Holter. Recording duration for both ECG Holter and CSF-3 device will be at least 7 minutes.
  Interventions: Device: CSF-3 watch, designed to monitor a user's heart rate based on ECG (electrocardiogram) and PPG (Photoplethysmograph) readings

INTERVENTIONS:
Device: CSF-3 watch, designed to monitor a user's heart rate based on ECG (electrocardiogram) and PPG (Photoplethysmograph) readings — The subjects will be connected to an ECG Holter, and an investigational Device will be placed simultaneously on the subject's wrist. All subjects in this phase will be asked to participate in a single continuous data recording measurement for seven (7) minutes
  Other Names: FDA cleared ECG Holter

SUMMARY:
CSF-3 is a wrist-worn medical device similar to a watch. It is designed to monitor a user's heart rate based on ECG (electrocardiogram) and PPG (Photoplethysmograph) readings, using off-the-shelf ECG and unique PPG chipsets with proprietary algorithms. ECG and PPG are the two primary technologies for measuring heart rate. ECG measures the bio-potential generated by electrical signals that control the expansion and contraction of heart chambers, while PPG uses light-based technology to sense the rate of blood flow as controlled by the heart's pumping action.

DETAILED DESCRIPTION:
The proposed clinical study is a prospective, open, single-center study to evaluate the performance and accuracy of the ECG and heart rate calculation of the CSF-3 investigational Device.

Subjects will be screened by the Principal Investigator. Subjects who meet the study's enrolment criteria will be recruited and fitted with an FDA cleared ECG Holter, and with the investigational Device (CSF-3).

At least 40 eligible subjects will be enrolled in a single center. Data collected from the subjects during the study will be included in the overall performance analysis of the ECG output. Subjects will perform an ECG and CSF-3 Device simultaneously Subjects will remain connected to both the ECG Holter and the CSF-3 Device at the study site for at least 7 minutes duration. The ECG and Holter will be stopped simultaneously. Both recordings data (ECG and CSF-3) will be uploaded and then synchronized offline using a dedicated and validated tool.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years old
* Able and willing to understand and sign the informed consent and follow instructions
* Screening ECG results of Sinus Rhythm
* Wrist size 14 cm (5.5"), Max 20 cm (7.8")

Exclusion Criteria:

* Subjects who are currently enrolled in other clinical investigation
* Subjects diagnosed with a cardiac disorder or any cardiac symptoms
* Subjects with SNR < 100
* Subjects with ECG quality range > 1 and < 30
* Individuals with electrical pacing by a pacemaker
* Subjects who are pregnant or breastfeeding
* Subjects with callous on the index finger or thumb (at fingerprint area)
* Subjects with active wound, prior soft tissue injury or skin conditions at the measurement location Sensitivity to the device material or ECG patches
* Subjects with tremors or otherwise unable to remain still for 15 minutes
* Subjects without two hands and sufficient fingers to complete the study
* Subjects unable to participate based upon investigator discretion

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
CSF-3 efficacy in ECG detection | 6 months
  Performance endpoint is defined as the ability of CSF-3 to detect beat-by beat Heart Rate in ECG signal with a sensitivity of no less than 96%, considering a false detection rate of not higher than 2%, and PPV of 80%.

SECONDARY OUTCOMES:
CSF-3 HR calculation | 6 months
  Performance endpoint is defined as the calculation of average Heart Rate with ARMS error<3BPM

CONTACTS AND LOCATIONS:
Locations (1):
- Fairview Health Services, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No